CLINICAL TRIAL: NCT03626948
Title: SK-1403 Long-term Treatment Study - Long-term Study in Patients With Secondary Hyperparathyroidism Receiving Hemodialysis -
Brief Title: SK-1403 Long-term Treatment Study; Long-term Study in Patients With Secondary Hyperparathyroidism Receiving Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJ1003
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SK-1403 (Experimental): Patients receive SK-1403 three times a week administered by intravenous bolus injection at the end of each hemodialysis for the whole treatment periods (52 weeks), with individual dose adjustment.
  Interventions: Drug: SK-1403

INTERVENTIONS:
Drug: SK-1403 — Patients receive SK-1403 three times a week administered by intravenous bolus injection at the end of each hemodialysis for the whole treatment periods (52 weeks), with individual dose adjustment.

SUMMARY:
To evaluate the safety and efficacy of treatment with SK-1403 for 52 weeks in patients with secondary hyperparathyroidism on maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Serum PTH>240 pg/mL at the screening
* Serum corrected Ca≥8.4 mg/dL at the screening
* Stable chronic kidney disease patients who undergo hemodialysis or hemodialysis filtration

Exclusion Criteria:

* Primary hyperparathyroidism
* Severe liver disease
* Severe cardiac disease
* History or family history of long QT syndrome
* Malignant tumor
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* A history of severe drug allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events or adverse drug reactions | 52 weeks
  Number of participants with adverse events or adverse drug reactions

SECONDARY OUTCOMES:
Rate of participants who achieved a serum iPTH level of ≥ 60 pg/mL and ≤ 240 pg/mL at each time point | 52 weeks
  Rate of participants who achieved a serum iPTH level of ≥ 60 pg/mL and ≤ 240 pg/mL at each time point; Assessed by laboratory test value
Measured values and Changes from baseline in serum PTH, Ca, ionized Ca, P, and serum Ca x P product | 52 weeks
  Measured values and Changes from baseline in serum PTH, Ca, ionized Ca, P, and serum Ca x P product; Assessed by laboratory test value

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site (there may be other sites in this country), Tokyo, Japan